| Study | Title: A More Physiological Feeding Process in |
|------------------|---------------------------------------------------|
| | Intermittent Infusion With Semi-solidification of |
| <u>nutrients</u> | <u>s</u> |
| Clinic | alTrails.gov ID: NCT 03017079 |
| Date: | 11/24/2016 |
| Respo | nsible party: Man Huang |
| Email | huangman@zju.edu.cn |

## **Statistical Analysis Plan**

Data were expressed as means ± standard deviations (SD) for quantitative variables and proportions for categorical and binary variables. Student's t test was used for statistical comparison between groups for continuous variables, general linear model for repeated measurement data, Fisher exact tests for categorical variables, and Mann-Whitney U test for ordinal variables. All tests for statistical significance were determined using an alpha level of 0.05. All analyses were performed using SPSS 17.0.